CLINICAL TRIAL: NCT02398617
Title: Facilitating End-Of-Life Decision Making and Preparedness Planning Among Heart Failure Patients Hospitalized for Advanced Disease
Brief Title: End-Of-Life Decision Making and Preparedness Planning Among Heart Failure Patients Hospitalized for Advanced Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment and need to refine protocol
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-192
Record Dates: First submitted 2015-02-20; First posted 2015-03-25 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; End of Life Care; Decision Making
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decision Making Intervention (Other): At their regularly scheduled admission follow-up visit with seven days of discharge, participants will be asked to bring their medical decision maker and participate in a semi-structured supplemental palliative care/education session facilitated by a heart failure nurse practitioner trained in palliative care discussions. Domains included in the intervention will include disease literacy and understanding, goals of care, legal issues for patients with terminal illness, symptom management, health-related quality of life, caregiver burden, patient autonomy, healthcare utilization, and establishment of end-of-life plans.
  Interventions: Other: Decision Making Intervention

INTERVENTIONS:
Other: Decision Making Intervention — At their regularly scheduled admission follow-up visit with seven days of discharge, participants will be asked to bring their medical decision maker and participate in a semi-structured supplemental palliative care/education session facilitated by a heart failure nurse practitioner trained in palliative care discussions. Domains included in the intervention will include disease literacy and understanding, goals of care, legal issues for patients with terminal illness, symptom management, health-related quality of life, caregiver burden, patient autonomy, healthcare utilization, and establishment of end-of-life plans.

SUMMARY:
Heart failure is a chronic and frequently terminal illness associated with poor quality of life and high burden of morbidity, re-hospitalization, and cost. Accordingly, recent guideline updates have highlighted the need for improved focus on end-of-life and palliative care of advanced heart failure patients, in whom symptom burden can be high and treatment options are often limited. The aims of this study are to evaluate the feasibility of implementing a semi-structured, outpatient, nurse practitioner-led, educational supportive care intervention concerning multiple domains of end-of-life care not often included in regular, outpatient clinic visits.

DETAILED DESCRIPTION:
This study will be a prospective pilot enrolling 10 patients with advanced disease admitted to the heart failure service at St. Luke's Mid America Heart Institute and who are not candidates for advanced therapies such as heart transplant or mechanical circulatory support (left ventricular assist device). Potential enrollees will be identified using a validated risk model that predicts death or poor quality of life in the six months after discharge from the hospital for heart failure exacerbation. Enrolled patients will complete validated questionnaires while still hospitalized, regarding health-related quality of life, illness acceptance, prioritization of different life goals, and confidence in decision-making regarding their terminal heart failure. Patients will then be given a paper exercise regarding delineation of an end-of-life plan and appointment of a surrogate medical decision-maker, to be completed after discharge. At their regularly scheduled admission follow-up visit with seven days of discharge, participants will be asked to bring their medical decision maker and participate in a semi-structured supplemental palliative care/education session facilitated by a heart failure nurse practitioner trained in palliative care discussions. Domains included in the intervention will include disease literacy and understanding, goals of care, legal issues for patients with terminal illness, symptom management, health-related quality of life, caregiver burden, patient autonomy, healthcare utilization, and establishment of end-of-life plans.

Outcomes to be measured after the intervention include repeated validated questionnaires and unstructured patient interviews at 1 month and, at 6 months, creation of a formalized end-of-life plan, change in code status, obtainment of an advanced directive, designation of a durable power of attorney, frequency of re-hospitalizations, emergency room visits and unscheduled clinic visits with providers, and death. These will be obtained at the time of regularly scheduled heart failure clinic follow-up visits or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* advanced heart failure
* ineligible for advanced therapies
* 50% risk of death or continued poor heart failure-related health status at 6 months from hospital discharge, based on validated risk score

Exclusion Criteria:

* Hospice enrollment
* Previous heart transplant or left ventricular assist device placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 month
  Heart failure-related quality of life
Decisional Conflict Scale | 1 month
  Decision-making confidence/readiness
Peace, Equanimity, and Acceptance in Cancer Experience (PEACE) Scale | 1 month
  Illness Acceptance
Kaldjian's Goals of Care at End of Life | 1 month
  Patient-ranked importance for different goals of care

SECONDARY OUTCOMES:
Death | 6 months
  Mortality
Code Status Change | 6 months
Advance Directive creation | 6 months
Durable Power of Attorney appointment | 6 months
Unscheduled Healthcare Encounter | 6 months
  Composite of re-hospitalizations, emergency department visits, urgent care visits, and unscheduled outpatient heart failure clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: John A Spertus, MD, MPH, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States